CLINICAL TRIAL: NCT03445312
Title: Safety and Effectiveness of a Laboratory Intervention to Effectively NOT Treat Asymptomatic Bacteriuria (SALIENT-A)
Brief Title: Safety and Effectiveness of a Laboratory Intervention to Effectively NOT Treat Asymptomatic Bacteriuria
Acronym: Salient
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Allison McGeer, Medical Director, Infection Prevention and Control, Mount Sinai Hospital, Canada
Other Study IDs: MSH 16-0302E
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Asymptomatic Bacteriuria; Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study cohort: All non-ICU medicine and surgery patients at Sinai Health System who have a mid-stream urine culture ordered
  Interventions: Behavioral: not processing urine cultures

INTERVENTIONS:
Behavioral: not processing urine cultures — microbiology lab will not process culture unless called

SUMMARY:
This is an observational cohort study of 1000 consecutive patients on medical and surgical wards at the Mount Sinai Hospital in Toronto who have a mid-stream urine culture ordered. When these cultures are ordered or received in the laboratory, a message is posted that the specimen will not be processed in the laboratory unless a call is received to say that the patient has local urinary symptoms. The goal is to establish whether not processing mid-stream urine cultures is safe.

DETAILED DESCRIPTION:
The clinical information system for Mount Sinai Hospital will be programmed such that, whenever a mid-stream urine sample is received in the microbiology laboratory from medical and surgical wards, the specimen will be held rather than processed. The system will reflex a result the specimen (either at a set time twice daily, or at the time the specimen is accessioned) with a message saying: "The great majority of positive urine cultures from inpatients without an indwelling urinary catheter represent asymptomatic bacteriuria and are no longer routinely processed. If you strongly suspect that your patient has developed a urinary tract infection or if you have mislabeled this specimen, please call the Microbiology laboratory within 48 hours to request processing of this urine culture".

Any urine being held in the microbiology laboratory will automatically generate an email alert to the study coordinator. Within 24 hours of receipt of the urine culture, the coordinator will confirm that the specimen was a midstream urine specimen, interview the patient, determine if they have had any symptoms of a urinary tract infection, and collect information on what other symptoms of infection were present when the culture was ordered, why the culture was ordered, and whether antibiotic therapy was started empirically.

All patients whose urines have not been processed will have a second follow-up visit/call at 72-96 hours to ensure that urinary symptoms have not developed or worsened. If symptoms develop/worsen, the study coordinator will have the investigator follow up.

All patients will have a follow-up telephone call/visit 28-35 days after the specimen is obtained to identify any intercurrent infections (including C. difficile infection), and any potential complications/adverse effects from antibiotics. Permission will be obtained to contact family or other attending physicians to clarify any information if necessary.

Data collected for each patient will include: age, gender, underlying medical conditions, reason for hospitalization, date of admission to hospital, service at admission and at the time urine specimen obtained, date urine specimen obtained, whether or not urine culture processed, urine culture results and date reported (if the urine culture was processed), urinalysis results (if ordered), why the urine culture was ordered, whether the patient had fever, hypothermia, dysuria, urgency, frequency, costophrenic angle tenderness, increased incontinence, presence/absence of delirium, presence/absence of any other behavior changes, whether the patient was capable of reporting urinary tract symptoms, duration of each symptom, whether or not empiric antibiotics were ordered (name, dose, duration) at the time the specimen was ordered and what the indication for antibiotics was, what the whether or not antibiotics ordered empirically were stopped if the urine culture was reported as negative; whether empiric antibiotics were appropriate to the pathogen (if the urine was cultured), whether the antibiotic regimen was changed in response to culture results (urine or other); what the final diagnosis from the most responsible physician was regarding the episode for which the urine culture was ordered; whether the episode met NHSN criteria for any infection, whether the patient developed any adverse events potentially associated with antibiotics (includes solicited: nausea, vomiting, diarrhea (including CDI), rash, vaginitis, any allergic reaction) and unsolicited - if the unsolicited are known to be adverse events associated with the antibiotic in question (eg. Stevens-Johnson syndrome with Septra, achilles tendon rupture with fluoroquinolones). Data will be collected by chart review, and by interview with the patient/next of kin.

For each patient in whom a serious adverse event occurs, a case summary will be prepared. Based on the case summary, hospital chart, and study notes, two internists/infectious disease physicians, otherwise unrelated to the study will be asked independently to assess whether the serious adverse event was associated with the failure to process a urine culture (if one was not processed), or associated with antibiotic prescribed for asymptomatic bacteruria. If the two physicians disagree, a third physician will review, and the three will meet to arrive at a consensus. If consensus cannot be achieved, the event will be recorded as associated with not performing the culture or with the antibiotic if 2 physicians of the 3 agree.

ELIGIBILITY:
Inclusion Criteria:

* inpatients on medical or surgical units at Mount Sinai Hospital

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All inpatients on medical and surgical units who have a mid-stream urine culture ordered
Sampling Method: Non-Probability Sample
Enrollment: 1394 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
serious adverse events (SAE) associated with not processing urine culture | 30 days
  serious adverse events associated with not processing urine culture

SECONDARY OUTCOMES:
Differences in SAE | 30 days
  Rate of serious adverse events in patients without symptoms who did and did not have urine specimens processed
SAE due to antibiotics | 30 days
  Rate of serious adverse events due to antibiotic therapy in patients who received antibiotics for asymptomatic bacteriuria
Non-response | 4 days
  Proportion of patients with symptomatic urinary tract infection (UTI) who did not respond to initial empiric antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Allison McGeer, Principal Investigator — Sinai Health System
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
individual patient data will not be available to other researchers. This is a quality improvement study